CLINICAL TRIAL: NCT01297348
Title: Postmarketing Study Of Lybrel In Relation To Venous Thromboembolism
Brief Title: Study Of Lybrel In Relation To Venous Thromboembolism
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Boston Collaborative Drug Surveillance Program (Other)
Responsible Party: Sponsor
Other Study IDs: 0858A2-4406; B3121004; NCT01316640 (obsolete NCT alias)
Record Dates: First submitted 2011-02-14; First posted 2011-02-16 (Estimated); Results first posted 2013-05-27 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-06

CONDITIONS: Venous Thrombosis; Pulmonary Embolism; Sinus Thrombosis, Intracranial
Keywords: Lybrel; levonorgestrel; ethinyl estradiol; venus thromboembolism (VTE); oral contraceptives (OC); safety; database study; case-control study
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Sinus Thrombosis, Intracranial | interventions — Levonorgestrel; Ethinyl Estradiol; lybrel; Ethinyl Estradiol-Norgestrel Combination; ethinyl estradiol, levonorgestrel drug combination; ovcon 35

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lybrel®: Current users of 90 ug levonorgestrel / 20 ug ethinyl estradiol - cases and controls (i.e., women diagnosed with new venus thromboembolism [VTE] and women not diagnosed with VTE).
  Interventions: Drug: 90ug levonorgestrel / 20 ug ethinyl estradiol
- Other OCs containing 20μg of ethinyl estradiol: Current users of oral contraceptives containing 20μg of ethinyl estradiol - cases and controls (i.e. women diagnosed with new VTE and women not diagnosed with VTE)
  Interventions: Drug: Oral Contraceptives containing 20 ug of ethinyl estradiol

INTERVENTIONS:
Drug: 90ug levonorgestrel / 20 ug ethinyl estradiol — This is a non-interventional observational database study, thus no interventions are offered to patients in the study.
  Other Names: Lybrel
  Groups: Lybrel®
Drug: Oral Contraceptives containing 20 ug of ethinyl estradiol — This is a non-interventional observational database study, thus no interventions are offered to patients in the study.
  Other Names: Lessina, Aviane, Junel 1/20, Junel FE 1/20, Levlite, Lutera, Alesse, Loestrin FE 1/20, Loestrin 1/20, Microgestin 1/20, Microgestin FE 1/20
  Groups: Other OCs containing 20μg of ethinyl estradiol

SUMMARY:
Lybrel® is an oral contraceptive that delivers low doses of levonorgestrel and ethinyl estradiol (90 μg/20 μg). Lybrel is taken on a continuous basis without a placebo or pill-free interval to inhibit menstrual cycle bleeding by delivering a steady level of the 2 hormones for as long as the drug is used. Lybrel was marketed in the US in July of 2007. The objective of this database case-control study is to estimate the risk of idiopathic VTE (deep vein thrombosis and pulmonary embolism) in current users of Lybrel (ethinyl estradiol 20ug/levonorgestrel 90ug) compared to current users of other oral contraceptives containing 20μg of ethinyl estradiol.

DETAILED DESCRIPTION:
The base population consists of all currently available data on current users (15-49 years old) of Lybrel and other oral contraceptives (OC) containing 20 µg ethinyl estradiol in the PharMetrics/IMS and MarketScan databases. From among the base population, the databases are then searched for any diagnosis of deep vein thrombosis (DVT), pulmonary embolism (PE), or cerebral venous sinus thrombosis (CVST) [referred to collectively as venous thromboembolism or VTE] that occurred after receipt of Lybrel or other oral contraceptives containing 20 µg ethinyl estradiol. The intent is to include newly diagnosed cases of VTE.

ELIGIBILITY:
Inclusion Criteria:

* New users of the study drugs (i.e., Lybrel and the comparison OCs)

Exclusion Criteria:

* No specific exclusion criteria for the base study cohort.

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The base population for each year of the study will comprise all 15 - 49 year old women who have any recorded prescriptions for either continuous use ethinyl estradiol 20ug/levonorgestrel 90ug or a cyclic oral contraceptive that contains 20 µg ethinyl estradiol. The women are identified from PharMetrics and MarketScan databases. Additionally, women are enrolled if the index prescription is a new one; this is defined as a prescription dispensed following a 4-month window in which no combined hormonal contraception prescriptions were filled.
Sampling Method: Non-Probability Sample
Enrollment: 598682 (Actual)
Dates: Start 2007-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0858A2-4406&StudyName=Study%20Of%20Lybrel%20In%20Relation%20To%20Venous%20Thromboembolism

RESULTS

PARTICIPANT FLOW:
Groups:
- Lybrel: Participants who were current or past users of Lybrel, a continuous use oral contraceptive containing levonorgestrel 90 microgram (mcg) and ethinyl estradiol 20 mcg, were observed.
- Other OCs: Ethinyl Estradiol 20 Mcg (EE-20): Participants who were current or past users of EE-20, cyclic oral contraceptives (OCs) containing ethinyl estradiol 20 mcg and a progestin, were observed.
Period: Overall Study
Arm/Group | Lybrel | Other OCs: Ethinyl Estradiol 20 Mcg (EE-20)
Started | 12281 | 586401
Completed | 12281 | 586401
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lybrel | Other OCs: Ethinyl Estradiol 20 Mcg (EE-20) | Total
Number analyzed (Participants) | 12281 | 586401 | 598682
Age, Customized [Number; unit: participants]
  15 to 19 years | 1549 | 151591 | 153140
  20 to 24 years | 1785 | 128757 | 130542
  25 to 29 years | 1925 | 99632 | 101557
  30 to 34 years | 2079 | 79184 | 81263
  35 to 39 years | 2074 | 56674 | 58748
  40 to 44 years | 1668 | 41299 | 42967
  45 to 49 years | 1201 | 29264 | 30465
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12281 | 586401 | 598682
  Male | 0 | 0 | 0
Percentage of Participants With Duration in Health Plan Before First Study OC Prescription [Number; unit: percentage of participants] — Duration in health plan was categorized into 4 categories: 6 to 12, 12 to 24, 24 to 60 and more than 60 months. Health plan was referred to the managed care plans which included information on paid claims for pharmaceuticals, medical diagnoses, procedures and demographic information on the participants.
  percentage of participants
    6 to 12 months | 27.6 | 24.0 | 51.6
    12 to 24 months | 39.1 | 31.9 | 71.0
    24 to 60 months | 27.5 | 37.0 | 64.5
    More than 60 months | 5.8 | 7.1 | 12.9
Percentage of Obese Participants [Number; unit: percentage of participants] | 3.7 | 3.0 | 6.7
Percentage of Participants With Gynecological Disorders [Number; unit: percentage of participants] — Percentage of participants were reported for following gynecological disorders: endometriosis, menstrual disorder and uterine leiomyoma.
  percentage of participants
    Endometriosis | 6.3 | 1.1 | 7.4
    Menstrual disorder | 26.8 | 24.8 | 51.6
    Uterine leiomyoma | 0.1 | 0.0 | 0.1
Percentage of Participants With Back Pain [Number; unit: percentage of participants] | 11.0 | 8.5 | 19.5
Percentage of Participants With Cardiovascular Disease [Number; unit: percentage of participants] | 3.3 | 2.8 | 6.1
Percentage of Participants With Hypertension [Number; unit: percentage of participants] | 6.3 | 3.7 | 10.0
Percentage of Participants With Hyperlipidemia [Number; unit: percentage of participants] | 8.9 | 5.5 | 14.4
Percentage of Participants With Diabetes [Number; unit: percentage of participants] | 2.2 | 1.7 | 3.9
Percentage of Participants With Asthma [Number; unit: percentage of participants] | 6.9 | 6.8 | 13.7
Percentage of Participants With Thyroid Disease [Number; unit: percentage of participants] | 0.8 | 0.8 | 1.6
Percentage of Participants With Length of Stay in Health Plan [Number; unit: percentage of participants] — Length of stay in health plan was categorized into: less than 1, 1 to 2, 3 to 4 and greater than or equal to 5 years. Health plan was referred to the managed care plans which included information on paid claims for pharmaceuticals, medical diagnoses, procedures and demographic information on the participants.
  percentage of participants
    Less than 1 year | 3.7 | 4.4 | 8.1
    1 to 2 years | 14.6 | 16.8 | 31.4
    3 to 4 years | 41.8 | 41.6 | 83.3
    Greater than or equal to 5 years | 40.0 | 37.2 | 77.2

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Idiopathic Venous Thromboembolism (VTE)
Description: Idiopathic VTE=deep vein thrombosis (DVT), pulmonary embolism (PE), or cerebral venous sinus thrombosis (CVST) occurring in absence of known risk factors. Incidence rate reported for current, past users. Current user=had claim for study OC prescription (Lybrel or other OCs containing ethinyl estradiol 20 mcg) whose filled use occurred within 30 days prior to or at index date. Past user=had claim for a study OC prescription whose filled use occurred between 90 to 31 days prior to index date. Index date=date of VTE diagnosis for case and corresponding date for matched control.
Time Frame: Index date (date of VTE diagnosis for case and corresponding date for matched control)
Population: Analysis population included all enrolled participants who met the eligibility criteria.
Measure: Number; unit: incidence rate per 100000 person-years
Groups:
- Other OCs: Levonorgestrel, Ethinyl Estradiol 20 Mcg (Levo-20): A subset of EE-20 group including participants who were current or past users of Levo-20, cyclic oral contraceptives (OCs) containing ethinyl estradiol 20 mcg and differing concentrations of levonorgestrel (progestin), were observed.
Arm/Group | Lybrel | Other OCs: Ethinyl Estradiol 20 Mcg (EE-20) | Other OCs: Levonorgestrel, Ethinyl Estradiol 20 Mcg (Levo-20)
Number analyzed (Participants) | 12281 | 586401 | 142860
incidence rate per 100000 person-years
  Current users | 176.2 | 87.5 | 50.5
  Past users | 54.1 | 18.0 | 17.6
Statistical Analysis 1: Comparison: Lybrel vs Other OCs: Ethinyl Estradiol 20 Mcg (EE-20); Incidence rate ratio (Lybrel/EE-20) along with corresponding 95 percent (%) confidence interval (CI) was reported for current users; Test type: Superiority or Other; Incidence rate ratio = 2.01, 95% CI 2-sided [1.23 to 3.29]
Statistical Analysis 2: Comparison: Lybrel vs Other OCs: Ethinyl Estradiol 20 Mcg (EE-20); Incidence rate ratio (Lybrel/EE-20) along with corresponding 95% CI was reported for past users; Test type: Superiority or Other; Incidence rate ratio = 2.99, 95% CI 2-sided [0.39 to 22.80]
Statistical Analysis 3: Comparison: Lybrel vs Other OCs: Levonorgestrel, Ethinyl Estradiol 20 Mcg (Levo-20); Incidence rate ratio (Lybrel/Levo-20) along with corresponding 95% CI was reported for current users; Test type: Superiority or Other; Incidence rate ratio = 3.49, 95% CI 2-sided [2.02 to 6.02]
Statistical Analysis 4: Comparison: Lybrel vs Other OCs: Levonorgestrel, Ethinyl Estradiol 20 Mcg (Levo-20); Incidence rate ratio (Lybrel/Levo-20) along with corresponding 95% CI was reported for past users; Test type: Superiority or Other; Incidence rate ratio = 3.07, 95% CI 2-sided [0.34 to 27.47]

2. Primary Outcome: Number of Idiopathic Venous Thromboembolism (VTE) Cases and Matched Controls
Description: Idiopathic VTE cases=new DVT, PE or CVST occurring in absence of known risk factors. Matched Control was defined as participants with no diagnosis of VTE matched for age, calendar time, exposure status and database. Current user=had claim for study OC prescription (Lybrel or other OCs containing ethinyl estradiol 20 mcg) whose filled use occurred within 30 days prior to or at index date. Past user=had claim for a study OC prescription whose filled use occurred between 90 to 31 days prior to index date. Index date=date of VTE diagnosis for case and corresponding date for matched control.
Time Frame: Index date (date of VTE diagnosis for case and corresponding date for matched control)
Population: Analysis population included all enrolled participants who met the eligibility criteria.
Measure: Number; unit: participants
Arm/Group | Lybrel | Other OCs: Ethinyl Estradiol 20 Mcg (EE-20) | Other OCs: Levonorgestrel, Ethinyl Estradiol 20 Mcg (Levo-20)
Number analyzed (Participants) | 12281 | 586401 | 142860
participants
  Current user: Case | 17 | 276 | 53
  Current user: Matched Control | 47 | 1144 | 254
  Past user: Case | 1 | 14 | 4
  Past user: Matched Control | 1 | 39 | 10
Statistical Analysis 1: Comparison: Lybrel vs Other OCs: Ethinyl Estradiol 20 Mcg (EE-20); Current user, case and matched control: Odds ratio (Lybrel/EE-20) and 95% CI were estimated using conditional logistic regression, conditional on matching factors (age, calendar time, exposure status and database); Test type: Superiority or Other; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.85 to 2.67]
Statistical Analysis 2: Comparison: Lybrel vs Other OCs: Levonorgestrel, Ethinyl Estradiol 20 Mcg (Levo-20); Current user, case and matched control: Odds ratio (Lybrel/Levo-20) and 95% CI were estimated using conditional logistic regression, conditional on matching factors (age, calendar time, exposure status and database); Test type: Superiority or Other; Odds Ratio (OR) = 2.53, 95% CI 2-sided [0.98 to 6.54]

ADVERSE EVENTS:
Description: The minimum criteria for reporting an adverse event (AE) (that is, identifiable participant, identifiable reporter, a suspect product, and event) were not available and adverse events were not reportable as individual AE reports in this observational non-interventional study.
Arm/Group | Lybrel | Other OCs: Ethinyl Estradiol 20 Mcg (EE-20)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Data for DVT, PE and CVST were not reported separately as the 3 were components of the primary endpoint VTE and not separate endpoints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.